CLINICAL TRIAL: NCT00614068
Title: Creating a Collaborative Field Research Organization
Brief Title: Effectiveness of Trauma-Focused Cognitive Behavioral Therapy in Treating Children With Post-Traumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 00-0996; R24MH063910 (NIH); DSIR SE-CE
Record Dates: First submitted 2008-02-11; First posted 2008-02-13 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Treatment; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Participants will receive 12 sessions of trauma-focused cognitive behavioral therapy over 3 months.
  Interventions: Behavioral: Trauma-focused cognitive behavioral therapy (TF-CBT)
- B (Active Comparator): Participants will receive 12 sessions of treatment as usual over 3 months.
  Interventions: Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Trauma-focused cognitive behavioral therapy (TF-CBT) — TF-CBT sessions will include trauma-focused treatment and will teach participants behavioral management and coping skills to overcome their PTSD.
  Arms: A
Behavioral: Treatment as usual (TAU) — TAU outpatient sessions will include routine community care and nontrauma-focused therapy.
  Arms: B

SUMMARY:
This study will compare the effectiveness of trauma-focused cognitive behavioral therapy versus standard care in treating children with post-traumatic stress disorder.

DETAILED DESCRIPTION:
Each year approximately 5 million children in the United States are exposed to some form of traumatic event, and nearly 40% of these children will go on to develop post-traumatic stress disorder (PTSD). There are a number of traumatic events that have been shown to cause PTSD in children, including natural disaster, physical or sexual abuse, loss of a loved one, and witnessing an act of violence. Children with PTSD may experience persistent generalized fear and anxiety, recurrent nightmares, mood swings, withdrawal, and depression. If left untreated, PTSD can cause serious distress for those affected, resulting in emotional, academic, and social problems. Trauma-focused cognitive behavioral therapy (TF-CBT), a form of psychotherapy that focuses on trauma, may be the most effective means of improving PTSD screening and treatment in community-based mental health services. Although TF-CBT has shown success in treating children with PTSD in the research setting, its use in community clinics remains limited. This study will compare the effectiveness of TF-CBT versus treatment as usual (TAU) in treating children with PTSD in community clinics. The study will also develop a community collaboration between a community mental health agency and an academic institution, both in New York City, to address childhood trauma and PTSD and to enhance research in community clinics.

Participation in this study will last about 3 months. Potential parent and child participants will first undergo initial assessments, which will include interviews and questionnaires concerning symptoms of PTSD. Eligible participants will then be assigned randomly to receive TF-CBT or TAU. Participants in both groups will attend 12 sessions over 3 months. TF-CBT sessions will include trauma-focused treatment and will teach participants behavioral management and coping skills to overcome their PTSD. TAU sessions will include routine community clinic care and will not involve a trauma-focused treatment component. Upon completion of treatment, participants will complete repeat interviews and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Seeking services at Jewish Board of Family and Children's Services outpatient clinics
* Meets DSM-IV criteria for PTSD
* Stable on medication for 1 month before study entry
* English-speaking

Exclusion Criteria:

* Active suicidality or anyone whose life circumstances might be considered peri-traumatic (e.g., active current abuse)
* Uncontrolled psychosis
* Severe mental retardation or severe brain damage
* Severe language comprehension barriers

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2007-01; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
University of California Los Angeles- Post-Traumatic Stress Disorder (UCLA-PTSD) Reaction Index | Measured at baseline and Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Claude M. Chemtob, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Rohini Luthra, PhD, Study Director — Icahn School of Medicine at Mount Sinai
Locations (8):
- United States (8):
  - Jewish Board of Family and Children's Services (Yeshiva Chanoch Lenaar), New York, New York
  - Jewish Board of Family and Children's Services (Staten Island), New York, New York
  - Jewish Board of Family and Children's Services (Beatman), New York, New York
  - Jewish Board of Family and Children's Services (Pelham), New York, New York
  - Jewish Board of Family and Children's Services (BoroPark), New York, New York
  - Jewish Board of Family and Children's Services (Break-Free Adolescent Services), New York, New York
  - Jewish Board of Family and Children's Services (South Brooklyn), New York, New York
  - Jewish Board of Family and Children's Services (Pride), New York, New York